CLINICAL TRIAL: NCT03081689
Title: Neo - Adjuvant Chemo / Immunotherapy for the Treatment of Resectable Stage IIIA Non Small Cell Lung Cancer (NSCLC): A Phase II Multicenter Exploratory Study
Brief Title: Neo-Adjuvant Immunotherapy With Nivolumab for Non Small Cell Lung Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP 16/03_NADIM
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Nivolumab 360 mg IV Q3W + Paclitaxel 200mg/m2 + Carboplatin AUC 6 IV Q3W in resectable stage IIIA N2-NSCLC adult patients followed by adjuvant treatment for 1 year with Nivolumab 240 mg IV Q2W for 4 months and Nivolumab 480mg Q4W for 8 months
  Interventions: Drug: Nivolumab 360 mg; Drug: Paclitaxel 200mg/m2; Drug: Carboplatin AUC 6

INTERVENTIONS:
Drug: Nivolumab 360 mg — Nivolumab 360 mg IV Q3W + Followed by adjuvant treatment for 1 year with Nivolumab 240 mg IV Q2W for 4 months and Nivolumab 480mg Q4W for 8 months
  Other Names: OPDIVO
Drug: Paclitaxel 200mg/m2 — Paclitaxel 200mg/m2 IV Q3W
  Other Names: Paclitaxel
Drug: Carboplatin AUC 6 — Carboplatin AUC 6 IV Q3W
  Other Names: Carboplatin

SUMMARY:
Phase II, single-arm, open-label multicenter study that assesses feasibility, safety and efficacy of combined neoadjuvant chemotherapy and immunotherapy with Nivolumab 360 mg IV Q3W + Paclitaxel 200mg/m2 + Carboplatin AUC 6 IV Q3W in resectable stage IIIA N2-NSCLC adult patients followed by adjuvant treatment for 1 year with Nivolumab 240 mg IV Q2W for 4 months and Nivolumab 480mg Q4W for 8 months.

DETAILED DESCRIPTION:
Phase II, single-arm, open-label multicenter study that assesses feasibility, safety and efficacy of combined neoadjuvant chemotherapy and immunotherapy with Nivolumab 360 mg IV Q3W + Paclitaxel 200mg/m2 + Carboplatin AUC 6 IV Q3W in resectable stage IIIA N2-NSCLC adult patients followed by adjuvant treatment for 1 year with Nivolumab 240 mg IV Q2W for 4 months and Nivolumab 480mg Q4W for 8 months.

Three cycles of neoadjuvant chemotherapy in combination with nivolumab will be administered.

After completion of neoadjuvant therapy (3 cycles) and before surgery, a tumor assessment will be done. Patients have to leave the study if there is evidence of progression. Patients with in-stable disease or partial response may be considered for surgery.

The report imaging response vs pathological response rate will be evaluated.

Patients eligible for the trial are those with a histological diagnosis or cytologically proven operable and resectable non-small-cell lung cancer. The total number of patients to be included will be 46 from 23 participating sites in Spain.

Accrual period of 1.5 years or until the inclusion of the last patient necessary to achieve the sample set in the protocol of 46 patients. After that all patients will be treated for 1 year with adjuvant immunotherapy and they will be followed during 3 years after adjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects eligible for the study are those with histologically- or cytologically- documented NSCLC who present stage IIIA disease. Locally advanced patients who present stage IIIA by the previous version can be included if are considered potencially resectable. In case of N2 disease suspicion, pathological assessment by EBUS, mediastinoscopy or thoracotomy has to be carried out for N2 confirmation.
2. Tumor should be considered resectable before study entry
3. Performance Status of 0 or 1
4. Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to registration/inclusion i. WBC ≥ 2000/μL ii. Neutrophils ≥ 1500/μL iii. Platelets ≥ 100 x103/μL iv. Hemoglobin > 9.0 g/dL v. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below): a. Female CrCl = (140 - age in years) x weight in kg x 0.85

1. 72 x serum creatinine in mg/dL

b. Male CrCl = (140 - age in years) x weight in kg x 1.00

1. 72 x serum creatinine in mg/dL vi. AST/ALT ≤ 3 x ULN vii. Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL) viii. INR/APTT within normal limits

   5. The patients need to have a forced expiratory volume (FEV1) ≥ 1.2 liters

   6. All patients are notified of the investigational nature of this study and signed a written informed consent in accordance with institutional and nacional guidelines, including the Declaration of Helsinki prior to any trial-related intervention.

   7. Patients aged > 18 years

   8. Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception.

   9. Women must not be breastfeeding

   10. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year.

   Exclusion Criteria:
   1. All patients carrying activating mutations in the TK domain of EGFR or any variety of alterations in the ALK gene.
   2. Patients with active, known or suspected autoimmune disease.
   3. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment.
   4. Patients with a history of interstitial lung disease cannot be included if they have sympthomatic ILD (Grade 3-4)
   5. Patients with other active malignancy requiring concurrent intervention
   6. Patients with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) are excluded unless a
   7. Any medical, mental or psychological condition which in the opinion of the investigator would not permit the patient to complete the study
   8. Patients who have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody,
   9. Patients with positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody)
   10. Patients with known history of testing positive for human immunodeficiency virus (HIV)
   11. Patients with history of allergy to study drug components excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Study Chair — spanish Lun Cancer Group
Locations (24):
- Spain (24):
  - Complejo hospitalario de la coruña, A Coruña, Coruña
  - Hospital Reina Sofía, Córdoba, Córdoba
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Vigo, Vigo, Pontevedra
  - Hospital de Cruces, Bilbao, Vizcaya
  - Hospital General de Alicante, Alicante
  - Hospital Universitari Quirón Dexeus, Barcelona
  - Hospital Universitari Vall Hebrón, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - H. Duran i Reynals-ICO, Barcelona
  - H. de la Princesa, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Fundación Jiménez Díaz, Madrid
  - H. La Paz, Madrid
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Clinico de Salamanca, Salamanca
  - Hospital Virgen de La Macrena, Seville
  - Hospital Virgen Del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - H. Gen. Univ. Valencia, Valencia
  - Hospital La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Provencio M, Serna-Blasco R, Nadal E, Insa A, Garcia-Campelo MR, Casal Rubio J, Domine M, Majem M, Rodriguez-Abreu D, Martinez-Marti A, De Castro Carpeno J, Cobo M, Lopez Vivanco G, Del Barco E, Bernabe Caro R, Vinolas N, Barneto Aranda I, Viteri S, Pereira E, Royuela A, Calvo V, Martin-Lopez J, Garcia-Garcia F, Casarrubios M, Franco F, Sanchez-Herrero E, Massuti B, Cruz-Bermudez A, Romero A. Overall Survival and Biomarker Analysis of Neoadjuvant Nivolumab Plus Chemotherapy in Operable Stage IIIA Non-Small-Cell Lung Cancer (NADIM phase II trial). J Clin Oncol. 2022 Sep 1;40(25):2924-2933. doi: 10.1200/JCO.21.02660. Epub 2022 May 16. PMID 35576508
- [Result] Provencio M, Nadal E, Insa A, Garcia-Campelo MR, Casal-Rubio J, Domine M, Majem M, Rodriguez-Abreu D, Martinez-Marti A, De Castro Carpeno J, Cobo M, Lopez Vivanco G, Del Barco E, Bernabe Caro R, Vinolas N, Barneto Aranda I, Viteri S, Pereira E, Royuela A, Casarrubios M, Salas Anton C, Parra ER, Wistuba I, Calvo V, Laza-Briviesca R, Romero A, Massuti B, Cruz-Bermudez A. Neoadjuvant chemotherapy and nivolumab in resectable non-small-cell lung cancer (NADIM): an open-label, multicentre, single-arm, phase 2 trial. Lancet Oncol. 2020 Nov;21(11):1413-1422. doi: 10.1016/S1470-2045(20)30453-8. Epub 2020 Sep 24. PMID 32979984
- [Derived] Provencio M, Nadal E, Insa A, Garcia Campelo R, Casal J, Domine M, Massuti B, Majem M, Rodriguez-Abreu D, Martinez-Marti A, de Castro J, Gomez de Antonio D, Macia I, Figueroa S, Fernandez Vago L, Calvo V, Palmero R, Sierra-Rodero B, Martinez-Toledo C, Molina-Alejandre M, Serna-Blasco R, Romero A, Cruz-Bermudez A. Perioperative chemotherapy and nivolumab in non-small-cell lung cancer (NADIM): 5-year clinical outcomes from a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2024 Nov;25(11):1453-1464. doi: 10.1016/S1470-2045(24)00498-4. Epub 2024 Oct 14. PMID 39419061
- [Derived] Sierra-Rodero B, Cruz-Bermudez A, Nadal E, Garitaonaindia Y, Insa A, Mosquera J, Casal-Rubio J, Domine M, Majem M, Rodriguez-Abreu D, Martinez-Marti A, De Castro Carpeno J, Cobo M, Lopez Vivanco G, Del Barco E, Bernabe Caro R, Vinolas N, Barneto Aranda I, Viteri S, Massuti B, Laza-Briviesca R, Casarrubios M, Garcia-Grande A, Romero A, Franco F, Provencio M. Clinical and molecular parameters associated to pneumonitis development in non-small-cell lung cancer patients receiving chemoimmunotherapy from NADIM trial. J Immunother Cancer. 2021 Aug;9(8):e002804. doi: 10.1136/jitc-2021-002804. PMID 34446577
- [Derived] Casarrubios M, Cruz-Bermudez A, Nadal E, Insa A, Garcia Campelo MDR, Lazaro M, Domine M, Majem M, Rodriguez-Abreu D, Martinez-Marti A, de Castro-Carpeno J, Cobo M, Lopez-Vivanco G, Del Barco E, Bernabe Caro R, Vinolas N, Barneto Aranda I, Viteri S, Massuti B, Barquin M, Laza-Briviesca R, Sierra-Rodero B, Parra ER, Sanchez-Espiridion B, Rocha P, Kadara H, Wistuba II, Romero A, Calvo V, Provencio M. Pretreatment Tissue TCR Repertoire Evenness Is Associated with Complete Pathologic Response in Patients with NSCLC Receiving Neoadjuvant Chemoimmunotherapy. Clin Cancer Res. 2021 Nov 1;27(21):5878-5890. doi: 10.1158/1078-0432.CCR-21-1200. Epub 2021 Aug 10. PMID 34376534
- [Derived] Laza-Briviesca R, Cruz-Bermudez A, Nadal E, Insa A, Garcia-Campelo MDR, Huidobro G, Domine M, Majem M, Rodriguez-Abreu D, Martinez-Marti A, De Castro Carpeno J, Cobo M, Lopez Vivanco G, Del Barco E, Bernabe Caro R, Vinolas N, Barneto Aranda I, Viteri S, Massuti B, Casarrubios M, Sierra-Rodero B, Tarin C, Garcia-Grande A, Haymaker C, Wistuba II, Romero A, Franco F, Provencio M. Blood biomarkers associated to complete pathological response on NSCLC patients treated with neoadjuvant chemoimmunotherapy included in NADIM clinical trial. Clin Transl Med. 2021 Jul;11(7):e491. doi: 10.1002/ctm2.491. PMID 34323406
- See also: Web page of the sponsor where users can find more information about SLCG studies — http://www.gecp.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 46
Age, Continuous [Median (Standard Deviation); unit: years] | 63.1 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 46
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Spain | 46
ECOG Performance Status Scale [Count of Participants; unit: Participants] — ECOG Performance Status Scale: It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability
  GRADES:
  ECOG 0: Fully active. ECOG 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours ECOG 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours ECOG 4: Completely disabled ECOG 5: Dead
  Participants
    ECOG 0 | 25
    ECOG 1 | 21
    ECOG 2 | 0
    ECOG 3 | 0
    ECOG 4 | 0
    ECOG 5 | 0
Cigarette Smoking History [Count of Participants; unit: Participants]
  Former smoker (≥ 1 year) | 25
  Current smoker | 21
  Never smoker | 0
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 26
  Squamous | 16
  NOS/Undifferenciated | 4
Tumor node, metastasis staging classification [Count of Participants; unit: Participants] — 8th ed.TNM for Lung Cancer Primary tumor (T) T0 means there is no evidence of a tumor T1-T4 describe the size & location of the tumor on a scale of 1 to 4. A larger tumor or a tumor that has grown deeper into nearby tissue will get a higher number Distant metastasis (M) M0:Cancer has not spread to other parts of the body M1:Cancer has spread to other parts of the body Regional lymph nodes (N) N1: Metastasis in ipsilateral peribronchial or ipsilateral hilar lymph & intrapulmonary nodes N2:Metastasis in ipsilateral mediastinal or subcarinal lymph node N3:Metastasis in contralateral node
  Participants
    T1N2M0 | 15
    T2N1M0 | 1
    T2N2M0 | 6
    T3N1M0 | 1
    T3N2M0 | 13
    T4N0M0 | 9
    T1N1M0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: The progression free survival is the percentage of the patients without disease progression
Time Frame: at 24 months from the first dose of neoadjuvant treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 46
percentage of participants | 77.1 [59.9 to 87.7]

2. Secondary Outcome: Overall Survival
Description: Percentage of patients are still alive
Time Frame: at 3 years from the first dose of neoadjuvant treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 46
percentage of participants | 89.9 [74.5 to 96.2]

ADVERSE EVENTS:
Time Frame: 40 months
Description: The severity of AE will be determined using CTCAE version 4.0
Arm/Group | Arm 1
All-Cause Mortality (participants affected / at risk) | 1/46
Serious Adverse Events (participants affected / at risk) | 3/46
Other Adverse Events (participants affected / at risk) | 43/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=46)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Increased lipase (Blood and lymphatic system disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=46)
Asthenia or fatigue (General disorders) | 23 (51)
Alopecia (Skin and subcutaneous tissue disorders) | 17 (17)
Nausea (Gastrointestinal disorders) | 15 (20)
Neurotoxicity (Nervous system disorders) | 13 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (19)
Diarrhoea (Gastrointestinal disorders) | 11 (18)
Skin disorders (rash) (Skin and subcutaneous tissue disorders) | 19 (40)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (14)
Vomiting (Gastrointestinal disorders) | 8 (12)
Decreased appetite or anorexia (General disorders) | 9 (16)
Constipation (General disorders) | 8 (12)
Paraesthesia (Nervous system disorders) | 8 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (20)
Anaemia (Blood and lymphatic system disorders) | 7 (7)
Increased aminotransferases (Blood and lymphatic system disorders) | 5 (5)
Increased serum amylase (Blood and lymphatic system disorders) | 3 (6)
Increased creatinine level (Blood and lymphatic system disorders) | 3 (3)
Increased lipase (Blood and lymphatic system disorders) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT03081689/Prot_SAP_000.pdf